CLINICAL TRIAL: NCT07066553
Title: Outcomes of Sepsis Patients in China: A Registry
Brief Title: Outcomes of Sepsis Patients in China (CHINA-SEP)
Acronym: CHINA-SEP
Status: Not yet recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Prof, Southeast University, China
Other Study IDs: 2025ZDSYLL251-P01
Record Dates: First submitted 2025-06-30; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Sepsis
Keywords: China; Sepsis; Intensive Care Unit; Outcomes
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis Group: The sepsis group comprised patients diagnosed with sepsis (Sepsis-3 criteria).

SUMMARY:
Sepsis poses a significant public health challenge in China. However, longitudinal real-world evidence on guideline adherence and patient outcomes remains scarce. This registry aims to address these gaps by systematically capturing guideline-concordant treatment patterns and associated outcomes in ICU patients diagnosed according to Sepsis-3.0 criteria across diverse settings, thereby generating actionable evidence to improve the quality of sepsis care nationwide.

DETAILED DESCRIPTION:
Sepsis is a major public health challenge in China and remains one of the leading causes of intensive care unit (ICU) admissions, accounting for approximately 20.6% of all ICU cases. However, longitudinal real-world data on adherence to clinical guidelines and associated patient outcomes remain limited. This multicenter observational registry is designed to systematically capture real-world management data from adult ICU patients diagnosed with sepsis according to Sepsis-3.0 criteria. The study will assess current treatment practices and document infection types, anatomical sites, pathogen profiles, and key clinical outcomes. By examining the relationship between treatment patterns and outcomes, this study aims to generate actionable evidence to improve the quality of sepsis care in China. The findings will help identify practice variability, support updates to national guidelines, and promote standardized, evidence-based management across the country.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged ≥18 years
* Sepsis diagnosis meeting Sepsis-3 criteria
* Informed consent signed by patient or legally authorized representative

Exclusion Criteria:

* Patients with a prior history of sepsis
* Sepsis diagnosis >48 hours prior to enrollment
* Current participation in clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sepsis (Sepsis-3 criteria) upon ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 5775 (Estimated)
Dates: Start 2025-07-18 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days after enrollment.

SECONDARY OUTCOMES:
Rate of compliance with sepsis bundle elements | Patient compliance with sepsis bundles will be assessed within 24 hours after ICU admission.
  This outcome quantifies the compliance rate, defined as the proportion of patients who completed all required sepsis bundle elements within the assigned 1-, 3-, or 6-hour window from time zero (time of sepsis recognition). Compliance rate is calculated as the number of patients who completed all clinically indicated bundle elements within the assigned time frame divided by the total number of eligible patients. The bundle elements include serum lactate measurement, blood culture collection prior to antibiotic administration, initiation of intravenous antibiotics, and administration of intravenous crystalloids for patients with hypotension or lactate levels greater than 4 mmol/L.
ICU mortality | From ICU admission to ICU discharge or death, up to 28 days
Ventilator-free days | 28 days after enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xie J, Wang H, Kang Y, Zhou L, Liu Z, Qin B, Ma X, Cao X, Chen D, Lu W, Yao C, Yu K, Yao X, Shang H, Qiu H, Yang Y; CHinese Epidemiological Study of Sepsis (CHESS) Study Investigators. The Epidemiology of Sepsis in Chinese ICUs: A National Cross-Sectional Survey. Crit Care Med. 2020 Mar;48(3):e209-e218. doi: 10.1097/CCM.0000000000004155. PMID 31804299
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338